CLINICAL TRIAL: NCT03427008
Title: mDOT: A Pilot Study of Video Directly Observed Therapy for Immunosuppressant Adherence in Adult Kidney Transplant Recipients
Brief Title: A Pilot Study of mDOT for Immunosuppressant Adherence in Adult Kidney Transplant Recipients
Acronym: mDOT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Merged IRB Created
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00164573
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-03

CONDITIONS: Medication Adherence; Transplant; Kidney
Keywords: mHealth; kidney transplantation; medication adherence; video directly observed therapy
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: This is a single center, prospective, randomized control trial with two arms. Participants in the intervention arm will use the mHealth app to manage and track their immunosuppression medical regimen post-transplant, and participants in the control arm will receive the current standard of follow-up care post-transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants in the control arm will be instructed to take their immunosuppressive medications as prescribed and attend required follow-up as is standard of care, and will not receive the mHealth app.
- mHealth Intervention (Experimental): Participants in the intervention arm will receive the mHealth app either while they are an inpatient post-transplant, or at their first post-transplant clinic visit. Study personnel will assist participants assigned to the mHealth intervention arm with downloading the mHealth app and explain its functioning. Participants will then use the application to aid in immunosuppressive medication adherence post-transplant.
  Interventions: Other: mHealth Intervention

INTERVENTIONS:
Other: mHealth Intervention — The mHealth app will allow transplant recipients to see their medication regimen, record themselves taking every dose, report side effects or symptoms, visualize their treatment progress, access educational content, and track appointments. This information is encrypted and transmitted to a HIPAA-secure web portal for providers to review.
  Arms: mHealth Intervention

SUMMARY:
The investigators are interested in whether or not the use of a mobile health (mHealth) application increases the rate of immunosuppression medication adherence among adult kidney transplant recipients. The investigators aim to test this by randomly assigning transplant recipients to the intervention (use of an mHealth app to manage and track their immunosuppression regimen) or control arm (standard of care) upon discharge from their initial transplant hospitalization, and tracking medication adherence over time. The study population will be approximately 50 adult kidney transplant recipients at the Johns Hopkins Hospital.

DETAILED DESCRIPTION:
In adult kidney transplant recipients, the leading predictor of rejection, kidney loss, and death is immunosuppressive medication nonadherence. An estimated one-third of kidney transplant recipients reportedly experience medication nonadherence, and even minor deviations from the required protocol have been shown to have negative effects. However, due to the lack of systematic measurements of adherence, the direct relationship between the level of immunosuppressive medication adherence and poor outcomes is not well understood. Therefore, the investigators believe that mHealth technologies could be a feasible way to allow clinicians and researchers to better understand baseline adherence measurements, and increase immunosuppression adherence among kidney transplant recipients.

We will use a mobile health platform that enables users to track dose-by-dose medication adherence through asynchronous, video directly observed therapy (DOT). This helps patients take their medication as prescribed and gives providers the assurance that their patients are supported and successful in treatment. DOT is the practice of watching a patient take every dose of medicine in-person, and has typically only been done in extreme cases because it can be both costly and burdensome: DOT is the standard of care for Tuberculosis treatment and has proven high-adherence rates. Through mHealth technology, DOT can be used more broadly and without added burden; emocha's technology allows this through enabling patients to use their mobile application to view their regimen, record themselves taking every dose of their medication, report side effects or symptoms, visualize their treatment progress, access educational content, and track appointments. This information is encrypted and transmitted to a HIPAA-secure web portal for providers to review. The aim of this study is to conduct a randomized control trial to compare medication adherence between patients who use the mHealth system against controls who do not.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥22 years)
* Receive a kidney transplant at the Johns Hopkins Hospital

Exclusion Criteria:

* Non-English speaking participants

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
12-week immunosuppression medication adherence | 12 weeks
  After 12 weeks in the study, patients will complete the 4-item immunosuppressant therapy adherence instrument (ITAS) to determine self-reported medication adherence (scores range from 0-12 with 0 indicating very poor adherence and 12 indicating perfect adherence). Additionally, immunosuppression level trends will be tracked via electronic medical record review to determine medication adherence.

SECONDARY OUTCOMES:
Feasibility of using the mHealth Application as Assessed by a Semi-Structured Interview and a 17-Item Survey | 12 weeks
  After 12 weeks in the study, participants will be asked to participate in a semi-structured phone interview in which they will answer questions regarding their medication adherence habits and their thoughts on how our mHealth technology was or was not helpful. They will also complete a 17-question post-satisfaction survey assessing their satisfaction levels with the mhealth technology. Responses in the 17-item survey are on a 7-item Likert scale, the range being Strongly Agree, Agree, Slightly Agree, Neither Agree nor Disagree, Slightly Disagree, Disagree, and Strongly Disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Macey Henderson, JD,PhD, Principal Investigator — Johns Hopkins University; Daniel Brennan, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Geest S, Borgermans L, Gemoets H, Abraham I, Vlaminck H, Evers G, Vanrenterghem Y. Incidence, determinants, and consequences of subclinical noncompliance with immunosuppressive therapy in renal transplant recipients. Transplantation. 1995 Feb 15;59(3):340-7. PMID 7871562
- [Background] Hong JH, Sumrani N, Delaney V, Davis R, Dibenedetto A, Butt KM. Causes of late renal allograft failure in the ciclosporin era. Nephron. 1992;62(3):272-9. doi: 10.1159/000187058. PMID 1436337
- [Background] Nevins TE, Kruse L, Skeans MA, Thomas W. The natural history of azathioprine compliance after renal transplantation. Kidney Int. 2001 Oct;60(4):1565-70. doi: 10.1046/j.1523-1755.2001.00961.x. PMID 11576374
- [Background] Shoskes DA, Avelino L, Barba L, Sender M. Patient death or renal graft loss within 3 yr of transplantation in a county hospital: importance of poor initial graft function. Clin Transplant. 1997 Dec;11(6):618-22. PMID 9408696
- [Background] Douglas S, Blixen C, Bartucci MR. Relationship between pretransplant noncompliance and posttransplant outcomes in renal transplant recipients. J Transpl Coord. 1996 Jun;6(2):53-8. doi: 10.7182/prtr.1.6.2.x11r325882657x21. PMID 9188358
- [Background] Desmyttere A, Dobbels F, Cleemput I, De Geest S. Noncompliance with immunosuppressive regimen in organ transplantation: is it worth worrying about? Acta Gastroenterol Belg. 2005 Jul-Sep;68(3):347-52. No abstract available. PMID 16268422
- [Background] Dew MA, DiMartini AF, De Vito Dabbs A, Myaskovsky L, Steel J, Unruh M, Switzer GE, Zomak R, Kormos RL, Greenhouse JB. Rates and risk factors for nonadherence to the medical regimen after adult solid organ transplantation. Transplantation. 2007 Apr 15;83(7):858-73. doi: 10.1097/01.tp.0000258599.65257.a6. PMID 17460556
- [Background] De Geest S, Sabate E. Adherence to long-term therapies: evidence for action. Eur J Cardiovasc Nurs. 2003 Dec;2(4):323. doi: 10.1016/S1474-5151(03)00091-4. No abstract available. PMID 14667488
- [Background] Gordon EJ, Gallant M, Sehgal AR, Conti D, Siminoff LA. Medication-taking among adult renal transplant recipients: barriers and strategies. Transpl Int. 2009 May;22(5):534-45. doi: 10.1111/j.1432-2277.2008.00827.x. Epub 2009 Jan 16. PMID 19175560
- [Background] De Geest S, Abraham I, Moons P, Vandeputte M, Van Cleemput J, Evers G, Daenen W, Vanhaecke J. Late acute rejection and subclinical noncompliance with cyclosporine therapy in heart transplant recipients. J Heart Lung Transplant. 1998 Sep;17(9):854-63. PMID 9773856
- [Background] Butler JA, Roderick P, Mullee M, Mason JC, Peveler RC. Frequency and impact of nonadherence to immunosuppressants after renal transplantation: a systematic review. Transplantation. 2004 Mar 15;77(5):769-76. doi: 10.1097/01.tp.0000110408.83054.88. PMID 15021846
- [Background] Takemoto SK, Pinsky BW, Schnitzler MA, Lentine KL, Willoughby LM, Burroughs TE, Bunnapradist S. A retrospective analysis of immunosuppression compliance, dose reduction and discontinuation in kidney transplant recipients. Am J Transplant. 2007 Dec;7(12):2704-11. doi: 10.1111/j.1600-6143.2007.01966.x. Epub 2007 Sep 14. PMID 17868065
- [Background] Chisholm MA, Lance CE, Williamson GM, Mulloy LL. Development and validation of the immunosuppressant therapy adherence instrument (ITAS). Patient Educ Couns. 2005 Oct;59(1):13-20. doi: 10.1016/j.pec.2004.09.003. PMID 16198214
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829